CLINICAL TRIAL: NCT01352780
Title: Psoriasis and Climate Therapy- Effect of Motivational Follow- up Calls on Clinical and Health Economic Parameters
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: OsloUHBHR
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2014-10

CONDITIONS: Psoriasis
Keywords: motivational interviewing; psoriasis; self management
MeSH Terms: conditions — Psoriasis | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- usual care (No Intervention): Motivational interviewing
  Interventions: Behavioral: Motivational interviewing

INTERVENTIONS:
Behavioral: Motivational interviewing — Motivational interviewing technique will be used to improve patient adherence to multiple health behaviour changes and support patients with psoriasis to self- manage effectively. The intervention will discuss on four main topics: diet, physical activity, stress management and psoriasis treatment.
  Motivational interviewing is a patient centered directive counselling technique that focuses on assisting patients to identify their problems and involves exploring ambivalence in an empathic manner. A key goal in motivational interviewing is to increase the importance of change from the client's perspective. This is accomplished by using specific types of open ended questions, selective reflections and reflective listening.

SUMMARY:
The aim of this study is to evaluate clinical and health economic parameters in relation to individual motivational counseling by phone.

DETAILED DESCRIPTION:
A chronic condition such as psoriasis requires a high level of self- management and requires for many patients behaviour change to improve health outcome. Changing behaviour is a challenge that requires a commitment by the patient to implement successfully. Motivational interviewing is a patient centered directive counseling technique that focuses on assisting patients to identify their problems and involves exploring ambivalence in an empathic manner. It is a well-known method of counseling, and is considered to be a useful intervention strategy in the treatment of lifestyle problems.

This study is a randomized controlled trial using telephone motivational interviewing. The counseling intervention comprises 6 telephone calls during a 12 week period, after attending 3 weeks of supervised climate therapy on the Canary Islands

ELIGIBILITY:
Inclusion Criteria:

* Conducted 3 weeks of supervised climate therapy in The Canary Islands
* Able to write and communicate in Norwegian
* PASI more than 7 on application

Exclusion Criteria:

* more than 5 climate therapy treatments during the last 10 years

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
SAPASI (+ PASI at T1 and T2) | Change in SAPASI from baseline, to 3 weeks, 6 weeks and 12 weeks
  The self-administered psoriasis area and severity index (SAPASI) is a structured instrument for measuring the severity of psoriasis.
HeiQ | change from baseline to 3 months, 6 months
  The heiQ™ is an Australian-developed health education impact evaluation system. It consists of a set of eight scales. Each scale is an independent questionnaire and together they provide a comprehensive profile of the intended outcomes of health education / self-management programs.

SECONDARY OUTCOMES:
15D | Change in 15D from baseline to 6 weeks and 12 weeks
  The 15D is a generic, comprehensive (15-dimensional), self-administered instrument for measuring HRQoL among adults (age 16+ years).
Questionnaire about lifestyle | Change in lifestyle parametres from baseline to 6 weeks and 12 weeks
  Questions about exercise, diet, stress, lifestyle change
BIPQ-2 | Change from baseline to 3 and 6 months
  short questionnaire about illness perception
Psoriasis Knowledge questionnaire | change in knowledge from baseline to 3 weeks, 3 months and 6 monthts
  40 questions about psoriasis and psoriasis treatment
Willingness to change to manage psoriasis | change from baseline to 3 months and 6 months
  8 questions about plans for change or conducted change managing psoriasis symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Astrid K. Wahl, PhD, Study Chair — University of Oslo, Departement of Health and Society,Department of Health Sciences
Locations (2):
- Norway (2):
  - Oslo University hospital, Department for clima therapy, Oslo, Oslo County
  - University of Oslo, Departement of health and society, Oslo

REFERENCES:
- See also: Related Info — http://www.med.uio.no/helsam/english/research/projects/psoriasis-climate-therapy/index.html